CLINICAL TRIAL: NCT03555760
Title: Observational Investigation of Patients' Readings of Pre-operative Informed Consent Forms
Brief Title: Patients' Readings of Pre-operative Informed Consent Forms
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Cagil Vural, Instructor, Ankara University
Other Study IDs: 08/07
Record Dates: First submitted 2018-05-22; First posted 2018-06-14 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Informed Consent; Awareness
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgery patient: Observation of informed consent form readings of all patients who are scheduled for surgery
  Interventions: Behavioral: Observation of informed consent form readings of all patients who are scheduled for surgery

INTERVENTIONS:
Behavioral: Observation of informed consent form readings of all patients who are scheduled for surgery — All patients who are scheduled for surgery will be observed for their initial reflex of inform consent form readings.

SUMMARY:
Patient informed consent is a form which contains the patient's probable outcome of the procedure to be performed, and the probable risk and benefit of the patient's knowledge of the illness. On the form, completely honest and detailed information based on the facts are shared with the patient. It will be beneficial to both the physician and the patient to make a correct and complete consent procedure. The view, feelings and thoughts including the continuous and mutual understanding effort between the patient individual and the follow-up health team (physician, nurse, etc.) are essential in this sense.

The information that must be provided covers all of the following:

* The health status of the patient and the diagnosis,
* The type of treatment proposed,
* The chances of success and duration,
* The risk that the treatment modality carries for the patient's health,
* The use of medicines and possible side effects,
* The consequences of the illness if the hospital does not accept the recommended treatment,
* Alternative treatment options and risks. The informed consent is different from the signing of the patient indicating that he approves the procedure to be performed. The main purpose is to provide information to the patient and to understand this knowledge. For this reason, before the signing of the proclamation, it is necessary to ensure that the patient is informed in accordance with his or her own cultural and educational level. In addition, the patient must be audited that he/she understands the given information.

The purpose of this study is to investigate whether the informed consent forms given to the patient after informing by the physician were read as the first reflex before signing.

ELIGIBILITY:
Inclusion Criteria:

* Being scheduled for surgery.
* Accept being part of the study and share information such as inform consent form readings and demographics.

Exclusion Criteria:

* Not to accept being part of the study and share information such as inform consent form readings and demographics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for surgery and legal guardian of patients under the age of 18.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Observations of patient readings of informed consent forms | 15 minutes
  Visual doctor observation of initial reflex of readings of informed consent forms before signing the documents. Outcome will be noted as positive or negative.
Patient demographics | Will be noted after outcome 1- 5 minutes
  Demographic features of patients recruited in the study will be noted, including age, gender, occupation and educational status.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Faculty of Dentistry, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided